CLINICAL TRIAL: NCT07160400
Title: A Phase 1 Clinical Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of IBI3032 After a Single Ascending Dose in Healthy Participants and After Multiple Ascending Doses in Participants With Overweight or Obesity
Brief Title: A Study of IBI3032 in Chinese Healthy Participants and Participants With Overweight or Obesity
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics Technology Limited (Shanghai R&D Center) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI3032A101
Record Dates: First submitted 2025-08-21; First posted 2025-09-08 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Part A: Healthy Part B: Overweight or Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single dose of IBI3032 administered orally. (Experimental): Part A
  Interventions: Drug: IBI3032 tablets
- Single dose of placebo administered orally. (Placebo Comparator): Part A
  Interventions: Drug: Placebo
- Multiple doses of IBI3032 administered orally. (Experimental): Part B
  Interventions: Drug: IBI3032 tablets
- Multiple doses of placebo administered orally. (Placebo Comparator): Part B
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Single dose placebo IBI3032 administered orally
  Arms: Multiple doses of placebo administered orally.; Single dose of placebo administered orally.
Drug: IBI3032 tablets — Single dose of IBI3032 administered orally
  Arms: Multiple doses of IBI3032 administered orally.; Single dose of IBI3032 administered orally.

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase 1 clinical study evaluating the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of a single ascending dose of IBI3032 in healthy participants and multiple ascending doses of IBI3032 in participants with overweight or obesity. It consists of 2 parts: Part A is a single ascending dose (SAD) study in healthy participants, and Part B is a multiple ascending dose (MAD) study in participants with overweight or obesity during the 4-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-65 years (inclusive) at the time of informed consent.
2. Participants must understand the procedures and methods of this study, be willing to complete the study in strict accordance with the clinical study protocol, and voluntarily sign the informed consent form.

Exclusion Criteria:

1. The investigator suspects that the participant may be allergic to any component of the study drug or GLP-1 receptor agonists, or have used GLP-1 receptor agonists within 3 months prior to screening.
2. History of diabetes, or HbA1c ≥ 6.5% and fasting blood glucose < 3.9 mmol/L or ≥ 7.0 mmol/Lat screening.
3. Presence of any other abnormalities in vital signs and laboratory tests that are clinically significant as judged by the investigator at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with adverse events (AEs) | Part A: Baseline up to Day 15
  An adverse event (AE) is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.
Number of Participants with adverse events (AEs) | Part B: Baseline up to Day 43
  An adverse event (AE) is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.
Number of Participants with One Serious Adverse Event(s) Considered by the Investigator to be Related to Study Drug | Part A: Baseline up to Day 15
  A summary of SAEs regardless of causality, will be reported in the Reported Adverse Events module.
Number of Participants with One Serious Adverse Event(s) Considered by the Investigator to be Related to Study Drug | Part B: Baseline up to Day 43
  A summary of SAEs regardless of causality, will be reported in the Reported Adverse Events module.
Number of Participants with More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug | Part A: Baseline up to Day 15
  A summary of other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module.
Number of Participants with More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug | Part B: Baseline up to Day 43
  A summary of other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module.

SECONDARY OUTCOMES:
Under the Serum Concentration-time Curve (AUC) of IBI3032 | Part A: Predose up to 168 hours postdose
  To evaluate the pharmacokinetic (PK) characteristics of a single dose of IBI3032 in healthy participants.
Under the Serum Concentration-time Curve (AUC) of IBI3032 | Part B: Predose up to 168 hours postdose
  To evaluate the pharmacokinetic (PK) characteristics of multiple doses of IBI3032 in participants with overweight or obesity.
maximum concentration (Cmax) of IBI3032 | Part A: Predose up to 168 hours postdose
  To evaluate the pharmacokinetic (PK) characteristics of a single dose of IBI3032 in healthy participants.
maximum concentration (Cmax) of IBI3032 | Part B: Predose up to 168 hours postdose
  To evaluate the pharmacokinetic (PK) characteristics of multiple doses of IBI3032 in participants with overweight or obesity.
time to maximum concentration (Tmax) of IBI3032 | Part A: Predose up to 168 hours postdose
  To evaluate the pharmacokinetic (PK) characteristics of a single dose of IBI3032 in healthy participants.
time to maximum concentration (Tmax) of IBI3032 | Part B: Predose up to 168 hours postdose
  To evaluate the pharmacokinetic (PK) characteristics of multiple doses of IBI3032 in participants with overweight or obesity.
clearance (CL) of IBI3032 | Part A: Predose up to 168 hours postdose
  To evaluate the pharmacokinetic (PK) characteristics of a single dose of IBI3032 in healthy participants.
clearance (CL) of IBI3032 | Part B: Predose up to 168 hours postdose
  To evaluate the pharmacokinetic (PK) characteristics of multiple doses of IBI3032 in participants with overweight or obesity.
apparent volume of distribution (V) of IBI3032 | Part A: Predose up to 168 hours postdose
  To evaluate the pharmacokinetic (PK) characteristics of a single dose of IBI3032 in healthy participants.
apparent volume of distribution (V) of IBI3032 | Part B: Predose up to 168 hours postdose
  To evaluate the pharmacokinetic (PK) characteristics of multiple doses of IBI3032 in participants with overweight or obesity.
elimination half-life (T1/2) of IBI3032 | Part A: Predose up to 168 hours postdose
  To evaluate the pharmacokinetic (PK) characteristics of a single dose of IBI3032 in healthy participants.
elimination half-life (T1/2) of IBI3032 | Part B: Predose up to 168 hours postdose
  To evaluate the pharmacokinetic (PK) characteristics of multiple doses of IBI3032 in participants with overweight or obesity.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality, China